CLINICAL TRIAL: NCT03208907
Title: An Open Label Randomized Comparative Study to Assess the Efficacy and Tolerability of Eurartesim® Versus Chloroquine and Nonrelapse Therapy With Primaquine for Uncomplicated Plasmodium Vivax Monoinfection Malaria
Brief Title: DHA-PQP vs Chloroquine and Primaquine for Radical Cure of Vivax Malaria in Brazil
Acronym: CuraVivax
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundação de Medicina Tropical Dr. Heitor Vieira Dourado (Other)
Collaborators: Ministry of Health, Brazil (Other Government); Oswaldo Cruz Foundation (Other)
Responsible Party: Principal Investigator, Wuelton Marcelo Monteiro, PhD, Director of Research, Fundação de Medicina Tropical Dr. Heitor Vieira Dourado
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 69476017.3.0000.0005
Record Dates: First submitted 2017-06-30; First posted 2017-07-06 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Malaria, Vivax; Therapeutics
Keywords: Vivax malaria; Radical cure; Elimination
MeSH Terms: conditions — Malaria, Vivax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CQ coadministered with PQ (Active Comparator): Chloroquine was administered for 3 days according to the brazilian protocol and Primaquine was administered for 14 days (0.50mg/kg/day)
  Interventions: Drug: CQ coadministered with PQ
- DHA-PQP coadministered with PQ (Experimental): Dihydroartemisinin/Piperaquine was administered according to the weight and Primaquine (0.50mg/kg/day)
  Interventions: Drug: DHA-PQP coadministered with PQ
- CQ and PQ starting on Day 42 (Experimental): Chloroquine was administered for 3 days according to the brazilian protocol and Primaquine started on Day 42 for 14 days (0.50mg/kg/day) [arm halted after preliminary analysis]
  Interventions: Drug: CQ and PQ starting on Day 42
- DHA-PQP and PQ starting on Day 42 (Experimental): Dihydroartemisinin/Piperaquine was administered for 3 days according to the weight and Primaquine started on Day 42 for 14 days (0.50mg/kg/day) [arm halted after preliminary analysis]
  Interventions: Drug: DHA-PQP and PQ starting on Day 42

INTERVENTIONS:
Drug: CQ coadministered with PQ — 113 subjects in a 3-day regimen treatment with the schizonticidal drug Chloroquine concomitantly to 14-day regimen treatment with Primaquine in a dose of 0.50 mg/kg/day.
  Other Names: Standard treatment with potential synergy
  Arms: CQ coadministered with PQ
Drug: DHA-PQP coadministered with PQ — In this treatment group, 112 subjects took DHA-PQP for three days and Primaquine for 14 days in the following dose: 0.50 mg/kg/day.
  Other Names: Experimental treatment with potential synergy
  Arms: DHA-PQP coadministered with PQ
Drug: CQ and PQ starting on Day 42 — 98 subjects in a 3-day regimen treatment with Chloroquine with a 14-day regimen treatment with Primaquine in a dose of 0.50 mg/kg/day starting on Day 42 after first dose of the schizonticidal drug.
  Other Names: Standard treatment with no potential synergy
  Arms: CQ and PQ starting on Day 42
Drug: DHA-PQP and PQ starting on Day 42 — 95 subjects in a 3-day regimen treatment with DHA-PQP with a 14-day regimen treatment with Primaquine in a dose of 0.50 mg/kg/day starting on Day 42 after first dose of the schizonticidal drug.
  Other Names: Experimental treatment with no potential synergy
  Arms: DHA-PQP and PQ starting on Day 42

SUMMARY:
Plasmodium vivax can be cause of severe malaria and mortality. There are serious public health implications associated with cases of P. vivax resistant to Chloroquine in the Americas as well there are efforts of many countries to eliminate this disease. In this way, it is critically important to evaluate an alternative radical cure treatment efficient to amazon scenario. The objectives of this trial are to demonstrate the superiority of adequate parasitological response at D42 of Dihydroartemisinin plus Piperaquine (DHA-PQP or Eurartesim®) versus Chloroquine and to evaluate the proportion of failure until D180 considering different starting days of Primaquine (0.50 mg/kg/day) for 14 days. It is an open, 4 arms, randomised, comparative trial. Total of 460 patients are initially planned to be included. To demonstrate the superiority of DHA-PQP compared to Chloroquine, the 95% confidence interval of the difference observed between both treatment success rates will be determined. Each recurrence will be passively and actively detected for 180 days.

DETAILED DESCRIPTION:
Dihydroartemisinin/Piperaquine (DHA-PQP or Eurartesim®) is recommended by World Health Organization Expert Board for the treatment of P.vivax malaria, in case of chloroquine-resistance (CQR). However, no clinical study has been conducted to assess the efficacy of DHA-PQP in P.vivax malaria in the Americas. According a study performed in Amazonas state, Brazil, Artesunate/Amodiaquine (ASAQ) exhibited high efficacy against CQ resistant Plasmodium vivax and is an adequate alternative in the study area. They recommend other studies with an efficacious comparator, longer follow-up and genotype-adjustment can improve CQR characterization. Other publication, a meta-analysis of randomized controlled trials, found nine publications from January 1989 to May 2013 in which DHA-PQP was more efficacious than CQ and Artemether/Lumefantrine in treating uncomplicated P. vivax malaria. However, this drug combination is not active against the hypnozoite stage of P. vivax. So, more efforts are required to establish how best combine this treatment with appropriate nonrelapse therapy.

In 2015, primaquine was assessed in high dose for 14 days as treatment for the hypnozoite forms with DHA-PQP or artesunate-pyronaridine (AS-PYR). Both the treatment arms offer evidence of good tolerability and efficacy.

In other previous study performed in an area with high chloroquine-resistance (Southern Papua, Indonesia), DHA-PQP was compared to ASAQ, but never compared to chloroquine by itself in areas where chloroquine still works. The objectives of this trial are to demonstrate the superiority of adequate parasitological response at D42 of Dihydroartemisinin plus Piperaquine versus Chloroquine and to evaluate the proportion of failure until D180 considering different starting days of Primaquine (0.50 mg/kg/day) for 14 days.

This clinical trial will be undertaken in the Amazonas State (Western Brazilian Amazon), in Manaus, at Fundação de Medicina Tropical Dr Heitor Vieira Dourado. The climate is tropical, with mean temperatures between 26°C and 30°C. It is a prospective, open-label, 4-arm, randomized and comparison trial. One hundred and fifteen (115) patients were planned to be enrolled in each treatment arm (after a preliminary analysis this number was increased to 184; total number of participants: 563). In this protocol, all the subjects will be screened to evaluate Glucose-6-phosphate dehydrogenase deficiency (G6PD) deficiency and the laboratorial tests (specially haemoglobin) in all the visits will be evaluated, as well. The referred deficiency is estimated to be 3% among men from the Amazon and essentially the A-type (african type), which leads to moderate deficiency and minor clinical complications. Each dose of the schizonticidal treatment will be administered by a study pharmacist, and the patient will be monitored for 30 minutes after administration. The assessment schedule will be done in days 1, 2, 3, 5, 7, 14, 21, 28, 42, 63, 90, 120, 150 and 180 (in addition, patient will be asked to come back to the health centre if fever occurs at any time).

ELIGIBILITY:
1 Inclusion criteria:

1. Adults and children over 6 months old (bodyweight>5 kg)
2. Body weight ≥5 kg and <100 kg (or above, upon justification of the investigator);
3. Biologically confirmed symptomatic Monoinfection by Plasmodium vivax, with parasite density between 100 and 100,000;
4. Efficient activity of the enzyme Glucose-6-Phosphate Dehydrogenase (G6PD);
5. Conditions for oral treatment;
6. Plans known to remain in the area of the research center during the follow-up period (180 days);
7. Hemoglobin concentration (Hb) at baseline> 7g / dL.
8. Women with reproductive potential (defined as women who are not in postmenopausal dust for at least 24 consecutive months, ie without menstruation within 24 months of admission to the study, and women who have not undergone surgical sterilization, specifically hysterectomy or bilateral oophorectomy) must have a negative pregnancy test or urine test within 48 hours prior to admission to the study; NOTE: The history reported by the participant is considered acceptable documentation of hysterectomy, bilateral oophorectomy, and menopause. Women are considered menopausal if they have not had a menstrual period for at least 12 months and have had a follicle-stimulating hormone (FSH) greater than 40 IU/L; if the FSH test not available, they must be in amenorrhea for 24 or more consecutive months. For women of child-bearing age, provision is made for using contraceptives as described in research product and primaquine information. Contraceptives should preferably be used at least two weeks prior to the start of study drug and continued for least one week after the discontinuation of any drug from the study. In case the patient reports that she has not used any contraceptive method in the two weeks prior to inclusion, she may be included if the doctor discards the possibility of pregnancy;
9. If the patient engage in sexual activity that could lead to pregnancy, women should use a form of contraception. At least one of the following methods should be used properly:

Condoms (male or female) with or without spermicidal agent; Diaphragm or cervical cap with spermicide Intrauterine device (IUD) Hormonal contraceptive Ligation Tubal microimplants i. Women with no reproductive potential, as defined above, are without the use of contraceptives.

j. Ability and willingness of the participant or legal guardian to provide free and informed consent in writing. Children who are able to understand the goals and risks of the study will sign a consent form.

2. Non-inclusion criteria:

a. Participate in another ongoing clinical trial; b. Signs of severe malaria such as: recent history of seizures (1-2 within 24 hours), unconscious state, lethargy, inability to drink or breastfeed, constant vomiting, inability to get up / sit due to weakness; c. Known hypersensitivity to any of the experimental medicinal products or to any of the excipients d. Evidence or report of ingestion of antimalarial treatment in the 60 days prior to inclusion; e. Concomitant or underlying serious illness, such as porphyria or psoriasis or known disturbances of electrolyte balance, such as hypokalemia or hypomagnesemia; f. Liver function test with ALT> 3x the reference value, which, according to the researcher's assessment, endangers the safety of the participant;

3. Exclusion criteria:

1. Withdrawal of consent;
2. The researcher's opinion, based on the risk and benefit assessment of the study;
3. Detection of mixed infection by malaria;
4. Women who become pregnant by the 63rd day of follow-up;
5. Women of childbearing age who give up using effective contraception during the first 63 days of follow-up study;
6. Discontinuation of blood schizonticidal treatment for any reason.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with negative parasitological test (schizonticidal therapy evaluation) | Day 42
  Schizonticidal efficacy will be assessed based on the absence of Vivax Plasmodium parasites in blood of the participants, confirmed by microscopy.
Number of participants with negative parasitological test (nonrelapse therapy evaluation) | Day 180
  Nonrelapse therapy efficacy will be assessed based on the absence of Vivax Plasmodium parasites in blood, confirmed by microscopy.

SECONDARY OUTCOMES:
Number of participants with negative parasitological test | 6 months (for this analysis will not be considered the primary outcomes dates (Day42 and D180)
  Therapy efficacy will be assessed based on the presence or absence of Vivax Plasmodium parasites in blood, confirmed by the presence or absence of parasites in peripheral blood by microscopy.
Number of participants with any biological intolerability | Until Day 28
  Evolution of haemoglobin levels until D28 will be monitored in all the scheduled visits and also on unscheduled visits.
Number of participants with any treatment-related adverse event of clinical tolerability | 6 months
  The participants will be clinically monitored. In all the scheduled visits a study physician will evaluate and register the clinical exam, and also obtain and update the clinical history to describe any adverse event. The participants will have also a card with a 24h phone number to contact in case of clinical symptoms or others needing.
Number of participants with treatment-related prolonged QT interval. | Day 3
  Electrocardiogram evaluation will be assessed after completion of schizonticidal treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marcus VG de Lacerda, MD, PhD, Principal Investigator — Fundação de Medicina Tropical Dr. Heitor Vieira Dourado
Locations (1):
- Fundação de Medicina Tropical Dr. Heitor Vieira Dourado, Manaus, Amazonas, Brazil

IPD SHARING:
Plan to Share IPD: Undecided